CLINICAL TRIAL: NCT01127165
Title: A Multi-center Comparative Trial of Low and High Dose Zonisamide in Children as Monotherapy
Brief Title: Low and High Dose Zonisamide in Children as Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2090-S082-404
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Results first posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2010-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zonisamide Low Dose Group (Experimental)
  Interventions: Drug: zonisamide low dose group
- Zonisamide High Dose group (Experimental)
  Interventions: Drug: zonisamide high dose group

INTERVENTIONS:
Drug: zonisamide low dose group — Initial dose was 2mg/kg/day, increased after 1~2 weeks to 3~4mg/kg/day.
  Arms: Zonisamide Low Dose Group
Drug: zonisamide high dose group — Initial dose was 2mg/kg/day, increased after 2~4 weeks to 6~8mg/kg/day.
  Arms: Zonisamide High Dose group

SUMMARY:
The purpose of this study is to confirm the adjustment dosage of zonisamide as monotherapy in children with epilepsy.

ELIGIBILITY:
Inclusion criteria:

1. Pediatric patients with epilepsy whose age is 2~15 years old.
2. Patients had at least two seizures for the last 6 months before entry.
3. Patients who had never taken antiepileptic drugs.
4. Patients with no chance of progressive disease based on the result of magnetic resonance imaging (MRI) or electroencephalogram (EEG).
5. Agreement of the guardian is needed.

Exclusion criteria:

1. Patients who have progressive central nervous system (CNS) disease.
2. Patients with serious disorder.
3. Patients who have abnormal liver function (serum glutamic oxaloacetic transaminase [SGOT]) or (serum glutamic pyruvic transaminase [SGPT]) values more than twice the normal values.
4. Patients who have abnormal renal function (blood urea nitrogen (BUN) or Creatinine) values more than three times the normal values.
5. Hemolytic anemia.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihee Mun, Study Director — Medical Department, Eisai Korea Inc.
Locations (11):
- South Korea (11):
  - Dongsan Medical Center of Keimyung Univ., Seoul
  - Gangnam Severance Hospital, Seoul
  - Inje Univ. Ilsan-Paik Hospital, Seoul
  - Inje Univ. Sanggye-Paik Hospital, Seoul
  - Korea Univ. Ansan Hospital, Seoul
  - Korea Univ. Guro Hospital, Seoul
  - National Health Insurance Corporation Ilsan Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang Univ. Cheonan Hospital, Seoul
  - Soonchunhyang Univ. Hospital, Seoul
  - Yeungnam University Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 11 centers in Korea during the period of March 2006 to July 2009.
Groups:
- Zonisamide Low Dose Group: Initial dose was 2 mg/kg/day, increased after 1~2 weeks to 3~4 mg/kg/day.
- Zonisamide High Dose Group: Initial dose was 2 mg/kg/day, increased after 2~4 weeks to 6~8 mg/kg/day.
Period: Overall Study
Arm/Group | Zonisamide Low Dose Group | Zonisamide High Dose Group
Started | 65 | 60
Completed | 49 | 41
Not Completed | 16 | 19
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 10 | 8
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide Low Dose Group | Zonisamide High Dose Group | Total
Number analyzed (Participants) | 65 | 60 | 125
Age Continuous [Mean (Standard Deviation); unit: years] | 8.3 (3.0) | 7.8 (3.0) | 8.1 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 26 | 60
  Male | 31 | 34 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 65 | 60 | 125
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Assessed As Seizure Free
Description: The percentage of participants who showed no seizure during the maintenance phase.
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Zonisamide Low Dose Group | Zonisamide High Dose Group
Number analyzed (Participants) | 49 | 41
percentage of participants | 63.1 | 57.6

2. Secondary Outcome: Change in Cognitive Assessment Korean-Wechsler Intelligence Scale for Children (K-WISC-Ⅲ)
Description: Cognitive assessment was performed using K-WISC-III. The total score of K-WISC-III is calculated as Full Scale IQ which ranges from 31 (worst) to 151(best). Higher scores indicate greater intelligence, lower scores indicate less intelligence. Thus a positive change indicated an improvement.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Zonisamide Low Dose Group | Zonisamide High Dose Group
Number analyzed (Participants) | 23 | 28
Scores on a Scale | -1.3913 (9.13) | 0.1071 (10.77)

3. Secondary Outcome: Change in Behavior Assessment Korea-Child Behavior Checklist (K-CBCL)
Description: The difference of K-CBCL between before and after the administration. K-CBCL is the Korean version of CBCL which is a standardized form that parents fill out to describe their children's behavioral and emotional problems. The total score ranges 0- 234, with higher scores indicating worse behavioral and emotional problems.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Zonisamide Low Dose Group | Zonisamide High Dose Group
Number analyzed (Participants) | 27 | 36
Scores on a Scale | -5.259 (7.31) | -1.611 (5.83)

4. Secondary Outcome: Change in Korean-Quality of Life Childhood Epilepsy (K-QOLCE)
Description: The difference of K-QOLCE between before and after the administration. K-QOLCE is Korean version of the Quality of Life in Childhood Epilepsy Questionnaire. The calculated total score ranges 0-100, with higher scores indicating higher quality of life.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Zonisamide Low Dose Group | Zonisamide High Dose Group
Number analyzed (Participants) | 23 | 28
Scores on a Scale | 4.7931 (0.167) | 1.2286 (0.776)

ADVERSE EVENTS:
Arm/Group | Zonisamide Low Dose Group | Zonisamide High Dose Group
Serious Adverse Events (participants affected / at risk) | 2/65 | 1/60
Other Adverse Events (participants affected / at risk) | 14/65 | 18/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide Low Dose Group (N=65) | Zonisamide High Dose Group (N=60)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute gastroenteritis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide Low Dose Group (N=65) | Zonisamide High Dose Group (N=60)
Somnolence (Psychiatric disorders) | 2 | 3
Dizziness (Nervous system disorders) | 1 | 3
Anorexia (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 2 | 1
Micturition Disorder (Renal and urinary disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 1
Weight Decrease (General disorders) | 2 | 0
Memory Impairment (Psychiatric disorders) | 1 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Sweating Decreased (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No